CLINICAL TRIAL: NCT04569734
Title: Safety and Feasibility of Intra-Cardiac Echocardiography in Guiding Left Atrial Appendage Occlusion With the Watchman Device: The ICE WATCHMAN Study (Data Coordinating Center)
Brief Title: The ICE WATCHMAN Trial
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mohamad Adnan Alkhouli, Principal Investigator, Mayo Clinic
Other Study IDs: 19-012524
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Left Atrial Appendage Closure With WATCHMAN Device Utilizing an Intra-procedural ICE Probe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Experimental: Treatment Group: Determination for participation in the study is based on institutional standard of care practice for assessment of WATCHMAN eligibility. Patients that are being considered for LAA Closure with WATCHMAN device implant based on a history of non-valvular atrial fibrillation who are at increased risk for stroke and systemic embolism based on CHADS2VASc score >2 but have an appropriate rationale to seek a non-pharmacologic alternative to anti-thrombotic therapy due to risks of anti-thrombotic therapy. Patients should be able to tolerate the WATCHMAN device implant procedure without the need for general anesthesia.
  Interventions: Procedure: WATCHMAN device implant procedure utilizing ICE probe

INTERVENTIONS:
Procedure: WATCHMAN device implant procedure utilizing ICE probe — The study will be a prospective, non-randomized multicenter registry of 100 patients undergoing LAA closure with the WATCHMAN device (possibly with WATCHMAN FLX when approved) utilizing an intra-procedural ICE probe under moderate sedation.
  Other Names: WATCHMAN

SUMMARY:
The aim of this multi-center study will be to assess the feasibility and safety of left atrial appendage (LAA) occlusion with the WATCHMAN™ device using a standardized intra-procedural intracardiac echocardiography (ICE) protocol under moderate sedation for procedural guidance. By eliminating the need for general anesthesia, the hope is to show a reduction in procedural time, decrease use of supplemental invasive procedures (central venous line, invasive arterial pressure monitoring and transesophageal echocardiography) and quicker patient recovery time. This approach can decrease healthcare resource utilization and safely simplify left atrial appendage closure with the WATCHMAN device.

DETAILED DESCRIPTION:
The study will be a prospective, non-randomized multicenter registry of 100 patients undergoing LAA closure with the WATCHMAN device (possibly with WATCHMAN FLX when approved) utilizing an intra-procedural ICE probe under moderate sedation. The primary feasibility endpoint will be ability to successfully implant the WATCHMAN device. Implant success is defined as confirmation of the device-specified release PASS (Position, Anchor, Size, Seal) criteria, successful device release, and adequate seal (defined as a residual leak <5 mm) as assessed by a core lab interpretation of the TEE 45 days post-implant. The primary safety endpoint will be a composite of major complications (major bleeding [intracranial bleeding, or bleeding requiring blood transfusion], pericardial effusion requiring pericardiocentesis or surgery, device embolization, procedural-related stroke, or procedural related death). Additional measured end points will be: freedom from conversion to general anesthesia and/or standard TEE during implant, the incidence and the size of iatrogenic atrial septal defect on 45 day TEE. The ICE procedural images will also be collected and analyzed by an independent committee composed of non-implanting interventionalist, and an imaging specialist. The images will be graded in quality as optimal (TEE equivalent), acceptable (adequate but not as detailed as TEE), and inadequate. This prospective study, along with its endpoints will be registered in clinicaltrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* The patients is eligible to undergo WATCHMAN device implant procedure
* The patient is eligible for short term anticoagulation therapy
* Ability to tolerate the procedure without the need for general anesthesia as assessed by the treating physician(s)
* Ability to give informed consent for the procedure
* The patient is able and willing to undergo the procedure under moderate sedation
* The patient is able and willing to return for required 45-day TEE.

Exclusion Criteria:

* Patient has contraindication for short term anticoagulation
* The patient has history of a hypercoagulable state per medical record documentation
* Pregnancy or planning to get pregnant during the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participation in the study is based on institutional standard of care practice for assessment of WATCHMAN eligibility. Patients that are being considered for LAA Closure with WATCHMAN device implant based on a history of non-valvular atrial fibrillation who are at increased risk for stroke and systemic embolism based on CHADS2VASc score >2 but have an appropriate rationale to seek a non-pharmacologic alternative to anti-thrombotic therapy due to risks of anti-thrombotic therapy. Patients should be able to tolerate the WATCHMAN device implant procedure without the need for general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Successfully implant the WATCHMAN device | 45 days post-implant
  Implant success is defined as confirmation of the device-specified release PASS (Position, Anchor, Size, Seal) criteria, successful device release, and adequate seal (defined as a residual leak <5 mm) as assessed by a core lab interpretation of the TEE 45 days post-implant
Absence of a composite of major complications | 7 days post-implant
  Absence of a composite of major complications such major bleeding [intracranial bleeding, or bleeding requiring blood transfusion], pericardial effusion requiring pericardiocentesis or surgery, device embolization, procedural-related stroke, or procedural related death)
Absence of a composite of major complications | 45 days post-implant
  Absence of a composite of major complications such major bleeding [intracranial bleeding, or bleeding requiring blood transfusion], pericardial effusion requiring pericardiocentesis or surgery, device embolization, procedural-related stroke, or procedural related death)

SECONDARY OUTCOMES:
Freedom from conversion to general anesthesia and/or standard TEE during implant | During procedure
  Freedom from conversion to general anesthesia and/or standard TEE during implant
Freedom from the incidence and the size of iatrogenic atrial septal defect | 45 days post-implant
  Freedom from the incidence and the size of iatrogenic atrial septal defect on 45 day TEE

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Adnan Alkhouli, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Pacific Heart Institute, Santa Monica, California
  - Mayo Clinic Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials